CLINICAL TRIAL: NCT00005663
Title: An International, Randomized, Double-Blind, Placebo-Controlled Study of Valacyclovir for the Suppression of Recurrent Ano-Genital HSV Infections in HIV-Infected Subjects
Brief Title: A Study of Valacyclovir as Treatment for Genital Herpes Simplex Virus in HIV-Infected Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 104C; HS230018
Record Dates: First submitted 2000-05-11; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-07

CONDITIONS: Herpes Simplex; HIV Infections; Herpes Genitalis
Keywords: Herpes Simplex; Antiviral Agents; Anus Diseases; Herpes Genitalis; Recurrence; valacyclovir
MeSH Terms: conditions — Herpes Simplex; HIV Infections; Herpes Genitalis; Anus Diseases; Recurrence | interventions — Valacyclovir

INTERVENTIONS:
Drug: Valacyclovir hydrochloride

SUMMARY:
The purpose of this study is to see if valacyclovir (Valtrex) is a safe and effective treatment for ano-genital HSV infections (herpes simplex virus infections of the anus and external genitals) in HIV-infected patients.

DETAILED DESCRIPTION:
Patients are randomized in a 2:1 ratio to receive either Valtrex or placebo, twice daily, for up to 6 months. Patients come to the clinic for routine monthly assessments for 6 months, and return to the clinic for evaluation within 24 hours of the first signs or symptoms of an ano-genital HSV recurrence. Once the clinician confirms the presence of at least the macular/papular lesion stage, double-blind suppressive therapy is discontinued and open-label treatment with a higher dose of Valtrex twice daily for 5 days is initiated. For the first recurrence, patients are instructed to return to the clinic for further clinical assessments on Day 5 of the recurrence. Patients who have not healed by Day 5 may be offered an additional five days of open-label treatment, as deemed appropriate by the clinical investigator. If an additional 5-day course of open-label treatment medication is dispensed, the patient returns to the clinic on Day 10 for evaluation. Patients who have not healed by Day 10 are managed as deemed appropriate by the investigator. Once treatment of the first ano-genital HSV recurrence is complete and the patient is healed, patients are switched to open-label suppressive therapy with Valtrex for the remainder of the study period (up to a maximum of 6 months). The total duration of the study for all patients is 6 months.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are at least 18 years old.
* Are HIV-positive.
* Have herpes simplex virus (HSV) 2.
* Have received combination anti-HIV therapy for at least 2 months before entering the study.
* Have had 4 or more recurrences of ano-genital HSV (herpes infection of the anus and genitals) in the last 12 months. (If patient is taking medication to control HSV, then he/she must have had 4 or more recurrences of ano-genital HSV per year before beginning regular anti-HSV therapy, which is defined as therapy of 12 or more weeks.)
* Agree to use effective methods of birth control from 2 weeks before taking study drug, throughout the study, and for 4 weeks after completing the study. (A female may be eligible if not able to have children.)

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have blood vessel disease.
* Are sensitive to acyclovir, Valtrex, famciclovir, or ganciclovir.
* Are unable to take medications by mouth.
* Have non-healed sores on the anus or genitals at beginning of study.
* Are using anti-herpes drugs. To be eligible for enrollment, patients currently using anti-herpes drugs must stop treatment with these drugs at the beginning of the study; however, therapy may be started again if the investigator finds it necessary.
* Are using interferon. Patients receiving interferon must stop interferon before beginning the study.
* Have kidney or liver problems.
* Are pregnant or breast-feeding.
* Have a type of HSV that is resistant to acyclovir, Valtrex, famciclovir, or ganciclovir.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-06

CONTACTS AND LOCATIONS:
Locations (24):
- United States (20):
  - East Bay AIDS Ctr, Berkeley, California
  - Pacific Oaks Research, Beverly Hills, California
  - Kraus Med Partners, Los Angeles, California
  - ViRx Inc, San Francisco, California
  - IDC Research Initiative, Altamonte Springs, Florida
  - Healthnet Institute, Fort Lauderdale, Florida
  - Univ of Miami School of Medicine, Miami, Florida
  - Treasure Coast Infectious Disease Consultants, Vero Beach, Florida
  - Palm Beach Research Ctr, West Palm Beach, Florida
  - Indiana Univ School of Medicine / Dept of Infect Dis, Indianapolis, Indiana
  - Univ of Minnesota, Minneapolis, Minnesota
  - Advanced Biomedical Research Inc, Hackensack, New Jersey
  - Nalle Clinic / Clinical Research Dept, Charlotte, North Carolina
  - Wake County Dept of Health, Raleigh, North Carolina
  - Westover Heights Clinic, Portland, Oregon
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Dr Alvan Fisher, Providence, Rhode Island
  - Baylor College of Medicine / Dept of Medicine, Houston, Texas
  - Richmond AIDS Consortium, Richmond, Virginia
  - Univ of Washington Virology Research Clinic, Seattle, Washington
- Canada (4):
  - Dr Barbara Romanowski, Edmonton, Alberta
  - Sunnybrook Health Science Ctr, Toronto, Ontario
  - Clinique Medicale L'Actuele, Montreal, Quebec
  - Centre De Recherche En Infectiologie, Ste Foy, Quebec